CLINICAL TRIAL: NCT05518552
Title: Effects of Manual Lumbar and Prone Traction on Clinical Variables in Patients With Non-specific Low Back Pain: A Randomized Control Study
Brief Title: Effects of Manual Lumbar and Prone Traction in Patients With Low Back Pain
Acronym: L&PtracinLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Obafemi Awolowo University (Other)
Responsible Party: Principal Investigator, Adesola Ojo Ojoawo, Principal Investigator, Obafemi Awolowo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ojo/2022/01
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Non-specific Low Back Pain
Keywords: Manual Lumbar Traction; Prone Traction; Pain Intensity; Low back pain; Disability
MeSH Terms: conditions — Pain; Low Back Pain

STUDY DESIGN:
Intervention Model Description: The group underwent manual lumbar traction with the patient lying prone on a couch using a manual technique by pulling from the ankles of the patient. Manual traction was performed by the therapist, pulling at the patient's ankles.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual Lumbar Traction (Experimental): The subjects consist of 25 patients with chronic low back pain. They underwent a manual lumbar traction with Physiotherapist pulling the patients while lying prone on a couch
  Interventions: Other: Manual lumbar traction
- Prone traction (Experimental): This group consist of patients with non specific chronic low back pain that were put on prone traction.
  Interventions: Other: Prone traction

INTERVENTIONS:
Other: Manual lumbar traction — Patient in the group were treated with manual traction
  Arms: manual Lumbar Traction
Other: Prone traction — Patient in the group were placed on prone traction
  Arms: Prone traction

SUMMARY:
The study determined the effects of manual Lumbar traction and prone traction on some clinical variables of patients with long standing low back pain.

DETAILED DESCRIPTION:
Traction therapy has been used in the management of low back pain (LBP) especially None Specific Low Back Pain. There are several recommendations on how lumbar traction should be performed, but the type of technique to be applied differs among the sources. Prone traction adapted from inversion therapy which is a form of gravitational traction has been reported to be effective in ameliorating disabilities of patients with low back pain as well reduce pain intensity. Manual lumbar traction is performed by the therapist, pulling at the patient's ankles and has been reported to be effective in relieving pain and reducing disability of patient with None Specific Low Back Pain (NSLBP). Documented evidences on the efficacy of traction in non-specific low back pain are still inconclusive. While manual lumbar traction seems more commonly used, probably owing to its positional advantage, its relative effectiveness compared with manual prone traction is still unknown, hence this study. Therefore, the aim of this study was to examine the efficacy of manual lumbar traction and prone traction on pain intensity, disability, spinal range of motion and quality of life in patients with None Specific Low Back Pain.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with Non-Specific Low Back Pain of not less than 3 months duration who were referred by a physician.
* Participants between the ages of 40 years and older.

Exclusion Criteria:

* Low back pain patients with specific pathology, such as systemic inflammatory diseases, pregnancy, fractures of the spine, tumors, infections.
* Participants with pathology affecting the trunk or upper and lower extremities

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
Visual Analogue scale | Change is being assessed at the Baseline, 3rd week and 6th week of treatment
  It measure pain intensity: 0 which is no pain to 10 which is excruciating pain

SECONDARY OUTCOMES:
Roland Morris low back pain Disability questionnaire | Change is being assessed at the Baseline, 3rd week and 6th week of treatment
  It measures the disability of the patients from 0, no disability to 24 which is the greatest disability
Goniometer | Change is being assessed at the Baseline, 3rd week and 6th week of treatment
  It measures spinal flexibility in "degree". The flexibility may start from 0 degree and the maximum depends on the flexibility of each participants

CONTACTS AND LOCATIONS:
Overall Officials: Adesola O Ojoawo, PhD, Principal Investigator — Obafemi Awolowo University Ile Ife
Locations (1):
- Obafemi Awolowo University, Ile-Ife, Osun State, Nigeria

IPD SHARING:
Plan to Share IPD: No
The data are kept with the principal investigator. Whosoever is interested can contact him for information

REFERENCES:
- [Background] Ostelo RW, de Vet HC, Knol DL, van den Brandt PA. 24-item Roland-Morris Disability Questionnaire was preferred out of six functional status questionnaires for post-lumbar disc surgery. J Clin Epidemiol. 2004 Mar;57(3):268-76. doi: 10.1016/j.jclinepi.2003.09.005. PMID 15066687
- [Background] Ozaktay AC, Cavanaugh JM, Asik I, DeLeo JA, Weinstein JN. Dorsal root sensitivity to interleukin-1 beta, interleukin-6 and tumor necrosis factor in rats. Eur Spine J. 2002 Oct;11(5):467-75. doi: 10.1007/s00586-002-0430-x. Epub 2002 Jun 4. PMID 12384756